CLINICAL TRIAL: NCT01738477
Title: Evaluation of Immunogenicity and Safety of GSK Biologicals' Tdap Booster Vaccine (Boostrix™) in Young Adults, Administered 10 Years After Previous Tdap Boosting
Brief Title: Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Boostrix™ Vaccine in Previously Boosted Young Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116570
Record Dates: First submitted 2012-11-21; First posted 2012-11-30 (Estimated); Results first posted 2017-12-27 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Tetanus; Acellular Pertussis; Diphtheria
Keywords: Booster; Tdap; Immunogenicity; Repeat dose; Safety; BoostrixTM; Persistence
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Boostrix

ARMS (2):
- Boostrix Group 2 (Experimental): Healthy male of female subjects, aged 19 to 30 years of age at the time of booster vaccination, who were randomized to the Lot A, Lot B or Lot C groups in study NCT00109330, received a second dose of Boostrix in this study.
  Interventions: Biological: Boostrix
- Boostrix Group 1 (Active Comparator): Healthy male of female subjects, aged 19 to 30 years of age at the time of booster vaccination, who received Massachusetts Public Health Biologic Laboratories combined tetanus and diphtheria vaccine in study NCT00109330, received the first dose of Boostrix in this study.
  Interventions: Biological: Boostrix

INTERVENTIONS:
Biological: Boostrix — Single dose intramuscular administration.

SUMMARY:
The purpose of this follow-up study is to evaluate the persistence of antibodies against all the vaccine antigens 10 years after booster vaccination with either Tdap or Td, and also to assess immunogenicity and safety of another dose of Boostrix, administered in this study. This protocol posting deals with objectives and outcome measures of the extension phase. The objectives and outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00109330).

DETAILED DESCRIPTION:
Subjects were previously vaccinated with either Boostrix or a control Td vaccine in study NCT00109330. Only subjects who were part of the primary study will be invited to participate in this study. All subjects will receive a single dose of Boostrix at Visit 1 (Day 0) and subjects will be observed till Visit 2 (Day 30) for safety in terms of solicited adverse events (during 4 days post vaccination), unsolicited adverse events (during 31 days post vaccination) and serious adverse event (during the trial period). A blood sample will be collected from all subjects before vaccination (Visit 1) and one month after vaccination (Visit 2) for antibodies estimation.

This summary has been updated following Protocol amendment 2 dated 03 October 2013. The protocol is being amended to facilitate enrolment by:

* - Extending the window period for re-vaccination from ± 6 months to ± 300 days from the Year 10 time point.
* - Extending the recruitment period from 6 months to 14 months. The format of non-inferiority criterion of the first co-primary objective has been updated to keep it aligned with the format of non-inferiority criterion of the second co-primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visit).
* Subjects who have received a dose of Tdap or Td vaccines 10 years (+/-300 days) back, in study NCT00109330.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the vaccine dose.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccine dose . For corticosteroids, this will mean prednisone (≥ 20 mg/day (for adult subjects), or equivalent. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 31 days after the dose of vaccine, with the exception of Influenza vaccine which is allowed throughout the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Previous vaccination against diphtheria, tetanus or pertussis since the last dose received in the Study NCT00109330.
* History of diphtheria, tetanus or pertussis diseases following the receipt of booster dose in the Study NCT00109330.
* Severe allergic reaction (e.g. anaphylaxis) after previous administration of any tetanus toxoid, diphtheria toxoid, or pertussis-antigen containing vaccines, or any component of Boostrix.
* Hypersensitivity to latex.
* Encephalopathy (e.g. coma, decreased level of consciousness, prolonged seizures) of unknown etiology occurring within 7 days following previous vaccination with pertussis-containing vaccine.
* History of any neurological disorders or seizures.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 99.5°F for oral, axillary or tympanic route, or ≥ 100.4°F for rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the booster dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions up to 1 month post-vaccination.

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2014-04-02 (Actual); Study Completion 2014-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- United States (19):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Woburn, Massachusetts
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, East Setauket, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Upper Saint Clair, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Started | 37 | 128
Completed | 36 | 124
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix Group 1 | Boostrix Group 2 | Total
Number analyzed (Participants) | 37 | 128 | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.3 (2.4) | 23.5 (2.1) | 23.5 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 57 | 75
  Male | 19 | 71 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1 | 6 | 7
  Oriental | 0 | 1 | 1
  Other | 5 | 7 | 12
  White/caucasian | 31 | 114 | 145

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T).
Description: A seroprotected subject was defined as a subject with anti-D/anti-T antibody concentrations above or equal (≥) to 0.1 IU/mL (international units per milliliter)
Time Frame: At Month 1
Population: The analysis was done on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, which included all evaluable subjects who had met the eligibility criteria, who complied with the procedures and intervals defined in the protocol and for whom assay results were available for antibodies against at least one study vaccine antigen.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 35 | 115
Participants
  Anti-D | 35 | 115
  Anti-T | 35 | 115
Statistical Analysis 1: Comparison: Boostrix Group 1 vs Boostrix Group 2; Non-inferiority in terms of seroprotection rates to diphtheria; Test type: Non-Inferiority — To assess the non-inferiority of the second dose of Boostrix (Boostrix 2 Group) minus first dose of Boostrix (Boostrix 1 Group) for anti-diphtheria. Objective of non-inferiority was considered to be met if the lower limit (LL) of the 95% confidence interval (CI) was greater than, or equal to -10%; Mean Difference (Final Values) = 0, 95% CI [-3.25 to 9.95]
Statistical Analysis 2: Comparison: Boostrix Group 1 vs Boostrix Group 2; Non-inferiority in terms of seroprotection rates to tetanus; Test type: Non-Inferiority — To assess the non-inferiority of the second dose of Boostrix (Boostrix 2 Group) minus first dose of Boostrix (Boostrix 1 Group) for anti-tetanus. Objective of non-inferiority was considered to be met if the LL of the 95% CI was above -10%; Mean Difference (Final Values) = 0, 95% CI [-3.25 to 9.95]

2. Primary Outcome: Antibody Concentrations Against Pertussis Toxoid (Anti-PT), Against Filamentous Hemagglutinin (Anti-FHA) and Against Pertactin (Anti-PRN).
Description: Concentrations were expressed in geometric mean concentrations (GMCs).
Time Frame: At Month 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 35 | 115
IU/mL
  anti-PT | 66.2 [50.8 to 86.2] | 87.3 [74.5 to 102.4]
  anti-FHA | 336.2 [250.0 to 452.2] | 290.5 [252.5 to 334.2]
  anti-PRN | 425.5 [281.9 to 642.3] | 463.3 [390.8 to 549.3]

3. Secondary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T).
Description: as for outcome 1
Time Frame: At Month 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 35 | 115
Participants
  Anti-D | 35 | 115
  Anti-T | 35 | 115

4. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Concentrations Above the Cut-off.
Description: The cut-off of the assay was ≥ 1.0 IU/mL.
Time Frame: At Month 0 and Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 35 | 115
Participants
  Anti-D at Month 0 | 23 | 70
  Anti-D at Month 1 | 34 | 115
  Anti-T at Month 0 | 27 | 86
  Anti-T at Month 1 | 35 | 115

5. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations.
Description: Concentrations were expressed as GMCs.
Time Frame: At Month 0 and Month 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 35 | 115
IU/mL
  Anti-D at Month 0 | 1.6 [1.1 to 2.3] | 1.6 [1.3 to 2.1]
  Anti-D at Month 1 | 6.8 [5.4 to 8.6] | 6.0 [5.3 to 6.9]
  Anti-T at Month 0 | 1.8 [1.4 to 2.4] | 1.8 [1.5 to 2.2]
  Anti-T at Month 1 | 9.9 [7.9 to 12.5] | 9.7 [8.5 to 11.0]

6. Secondary Outcome: Antibody Concentrations Against Pertussis Toxoid (Anti-PT), Against Filamentous Hemagglutinin (Anti-FHA) and Against Pertactin (Anti-PRN).
Description: Concentrations were expressed in geometric mean concentrations (GMCs).
Time Frame: At Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 35 | 115
IU/mL
  anti-PT | 5.3 [3.4 to 8.2] | 9.9 [8.1 to 12.2]
  anti-FHA | 21.7 [13.4 to 35.4] | 36.9 [31.5 to 43.3]
  anti-PRN | 27.8 [13.7 to 56.3] | 71.6 [56.7 to 90.6]

7. Secondary Outcome: Number of Subjects With a Booster Response to Anti-D and Anti-T.
Description: Booster response to anti-D and anti-T antigens was defined as:
  * for initially seronegative subjects with pre-booster antibody concentration below 0.1 IU/mL, an increase of at least four times 0.1 IU/mL one month after vaccination,
  * for initially seropositive subjects with pre-booster antibody concentration ≥ 0.1 IU/mL, an increase of at least four times the pre-booster antibody concentration one month after vaccination.
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 35 | 115
Participants
  Anti-D | 14 | 47
  Anti-T | 21 | 64

8. Secondary Outcome: Number of Subjects With a Booster Response to Anti-PT, Anti-FHA and Anti-PRN.
Description: Booster response to pertussis antigens was defined as:
  * for initially seronegative subjects (pre-booster antibody concentration below the assay cut-off) with an increase of at least four times the assay cut-off one month after vaccination;
  * for initially seropositive subjects with anti-body concentration < four times the assay cut-off with an increase of at least four times the pre-booster antibody concentration one month after vaccination;
  * for initially seropositive subjects with anti-body concentration ≥ four times the assay cut-off with an increase of at least two times the pre-booster antibody concentration one month after vaccination.
Time Frame: At Month 1.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 35 | 115
Participants
  Anti-PT | 33 | 106
  Anti-FHA | 34 | 104
  Anti-PRN | 29 | 79

9. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: The solicited local symptoms assessed were Pain, Redness and Swelling. Any = any solicited local symptom regardless of intensity.
Time Frame: During the 4 days (Day 0 - 3) follow-up period after vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with a study vaccine administration dose documented and the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Groups:
- Boostrix Group 1: Healthy male of female subjects, aged 19 to 30 years of age at the time of booster vaccination, who received Massachusetts Public Health Biologic Laboratories combined tetanus and diphtheria vaccine in study NCT00109330, received the first dose of Boostrix™ in this study.
- Boostrix Group 2: Healthy male of female subjects, aged 19 to 30 years of age at the time of booster vaccination, who were randomized to the Lot A, Lot B or Lot C groups in study NCT00109330, received a second dose of Boostrix™ in this study.
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 36 | 125
Participants
  Any Pain | 21 | 97
  Any Redness | 15 | 47
  Any Swelling | 7 | 30

10. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: The solicited local symptoms assessed were Fatigue, Gastrointestinal, Headache and Fever. Any = any solicited general symptom regardless of intensity.
Time Frame: During the 4 days (Day 0 - 3) follow-up period after vaccination.
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 36 | 125
Participants
  Any Fatigue | 8 | 38
  Any Gastrointestinal Symptoms | 1 | 11
  Any Headache | 8 | 40
  Any Fever | 1 | 3

11. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an adverse event (AE) reported in addition to those solicited during the clinical study. Any solicited symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: During the 31 days (Day 0 - 30) after vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with a study vaccine administration dose documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 37 | 128
Participants | 10 | 33

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to 31 days post-vaccination.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group 1 | Boostrix Group 2
Number analyzed (Participants) | 37 | 128
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 4-days (Days 0-3) post-vaccination period; Unsolicited AE(s): during the 31-day (Days 0-30) post-vaccination period; SAE(s): from Month 0 to Month 1.
Arm/Group | Boostrix Group 1 | Boostrix Group 2
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/128
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/128
Other Adverse Events (participants affected / at risk) | 30/37 | 107/128
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix Group 1 (N=37) | Boostrix Group 2 (N=128)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 15 (15) | 47 (47)
Fatigue (General disorders) | 8 (8) | 38 (38)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 11 (11)
Headache (Nervous system disorders) | 11 (15) | 46 (56)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 21 (21) | 97 (97)
Swelling (General disorders) | 7 (7) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.